CLINICAL TRIAL: NCT00565227
Title: A Phase I Study of Suberoylanilide Hydroxamic Acid (Vorinostat) (NSC 701852) in Combination With Docetaxel in Patients With Advanced and Relapsed Solid Malignancies
Brief Title: Phase I Study of Vorinostat in Combination With Docetaxel in Patients With Advanced and Relapsed Solid Malignancies.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: closed due to toxicity
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2006.026
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Non-Small-Cell Lung Carcinoma; Prostate Cancer; Bladder Cancer; Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms; Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Vorinostat; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- docetaxel plus vorinostat (Experimental)
  Interventions: Drug: vorinostat (suberoylanilide hydroxamic acid); Drug: docetaxel

INTERVENTIONS:
Drug: vorinostat (suberoylanilide hydroxamic acid) — Vorinostat will be administered by mouth as a pill for the first 14 days on a continuous basis during of each 21-day cycle (2 weeks of treatment, 1 week break).
  Other Names: Zolinza,NSC 701852
Drug: docetaxel — Docetaxel will be administered as an intravenous infusion (through the vein) on day 4 of each 21-day cycle.
  Other Names: Taxotere

SUMMARY:
Vorinostat (Suberoylanilide Hydroxamic Acid; NSC 701852) is a drug that inhibits an enzyme that plays a key role in the regulation of cell survival, growth, and eventual cell death, all of which play a role in cancer. As a result, this drug has the potential to affect a tumor's ability to survive. Vorinostat is the most potent drug of its kind that is currently under investigation in clinical trials. The primary objective of this study is to define the maximum safest dose of vorinostat in combination with a standard chemotherapy agent, docetaxel, in patients with advanced and relapsed lung, bladder, or prostate cancer.

DETAILED DESCRIPTION:
Vorinostat (also known as Suberoylanilide Hydroxamic Acid) is a new investigational drug that is not approved by the Food and Drug Administration. This drug has shown promising activity against a number of cancers. We want to determine if treatment with vorinostat in combination with a standard type of chemotherapy (docetaxel [Taxotere™]) is safe and possibly better than treatment with docetaxel alone. We also want to find out more about how patients and the cancer will react to the drugs, what happens to vorinostat in the human body (how your body reacts to this drug and breaks it down) and about its side effects when used in combination with chemotherapy (docetaxel).

The purpose of this study is to:

* Test the safety of the research study drug, vorinostat
* To determine if any toxicities or severe side effects occur when combining vorinostat with docetaxel (a standard chemotherapy treatment)
* To study how your body takes in, breaks down and responds to vorinostat
* To obtain more evidence of the ability of vorinostat to react against cancer, such as the kind that you have.

The use of vorinostat in combination with chemotherapy such as docetaxel may result in improved response of the cancer to treatment. Indeed, vorinostat may have an added benefit with docetaxel by promoting cancer cell death. This is because both drugs can interfere with the ability of the cancer to grow, although the way vorinostat does this is not clearly defined. Vorinostat and docetaxel both can disrupt the cancer's ability to produce daughter cancer cells and therefore, the administration of vorinostat before docetaxel is hoped to be better then either drug alone.

ELIGIBILITY:
Inclusion Criteria:

1. There is no limit on prior courses of chemotherapy as long as the regimen did not contain docetaxel. Prior use of paclitaxel (Taxol) or other taxanes is permissible.
2. Only patients with non-small cell lung, prostate, and bladder/urothelial cancer that has progressed after chemotherapy or after hormone therapy.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 3 weeks.
2. Patients may not be receiving any other investigational agents nor had prior treatment with histone deacetylase (HDAC) inhibitors (i.e. Valproic acid, PXD-001, Depsipeptide, MS-275 and LAQ-824)
3. Significant cardiovascular disease including congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-04; Primary Completion 2008-11 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The TITE-CRM dose escalation scheme will be used in this study to determine the maximum tolerated dose (MTD) of the combination therapy. | After 25 evaluable patients are accrued, a final set of side-effect estimates will be produced for each dose level, and the MTD will be the highest dose with a side-effect estimate at or below the target toxicity estimate of 30%.

SECONDARY OUTCOMES:
Although response is not the primary endpoint of this trial, patients with measurable disease will be assessed by standard criteria. | For the purposes of this study, tumor response will be assessed every 6 weeks.
To evaluate the blood levels of vorinostat and docetaxel when administered in combination. | All blood levels of the drugs will be conducted during the first cycle of chemotherapy only.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Bradley, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States